CLINICAL TRIAL: NCT02865759
Title: Empowering Women to Shorten Pre-hospital Delay After Decreased Fetal Movements and Simultaneously Lower the Frequency of Unwarranted Visits - a Randomized Study
Brief Title: Mindfetalness to Improve Pregnancy Outcome
Acronym: Mindfetal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sophiahemmet University (Other)
Collaborators: Karolinska Institutet (Other); Göteborg University (Other)
Responsible Party: Principal Investigator, Ingela Radestad, Principal Investigator, Sophiahemmet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-2
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Pregnancy Outcomes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfetalness (Experimental): The pregnant woman will be informed about the possibility of practicing Mindfetalness verbally, in a brochure and at a website. The practice is described as spending 15 minutes every day from gestational week 28 to get to know the fetal movement pattern. The fetus must be awake when she practice Mindfetalness and the woman is suggested to lay on her left side when she observe the fetal movements. In the brochure as well at the website the woman can write down something about the nature, frequency or strength of the fetal movements. If the woman experiences decreased frequency of fetal movements or weaker movements she is instructed to seek health-care without unnecessary delay.
  Interventions: Behavioral: Mindfetalness
- Routine Care (No Intervention): No activities will take place in the antenatal clinics randomized to routine care.

INTERVENTIONS:
Behavioral: Mindfetalness — The pregnant woman is motivated to practice Mindfetalness verbally, by a brochure and at a website.
  Arms: Mindfetalness

SUMMARY:
To improve pregnancy outcome, 39 000 pregnant women will be randomized to receive information about Mindfetalness or to routine care. The level of randomization will be the antenatal clinics in the Stockholm area.

DETAILED DESCRIPTION:
The investigators have randomized 33 antenatal clinics in Stockholm to the intervention (receiving information about Mindfetalness) and 30 to routine care. The randomization was performed in blocks according to varying yearly volumes of pregnant women and socio-economic residential area. Three small clinics, with a total of 85 women listed in 2015, were not randomized. Another four clinics, receiving referrals of women with need for specialized care, were not randomized either. The recruitment is restricted to the 63 randomized clinics. In a pilot study in one antenatal clinic, the intervention has been tested among 102 women. A run-in period will start at high-volume antenatal clinics 1 September 2016, one month before the investigators start to register the women that will be observed for pregnancy outcome. All information, including that of possible effect-modifying and possible confounding factors, will be fetched from population-based registers and linked by the personal identify number unique for each resident in Sweden. The Swedish Medical Birth Register, Obstetrix, the Swedish Educational Register, the Prescribed Drug Register and the National Patient Register provide the information. By this design, and the analyses according to the intention-to treat principle, attrition and differential misclassification of outcome becomes negligible. Non-differential misclassification of the predictor (Mindfetalness or no Mindfetalness) will be substantial, diluting the effect estimates. This dilution may be compensated by the large size of the trial. Since the unit of randomization is the antenatal clinics residual confounding is an issue. The investigators will have, however, information on important possible confounding factors, including educational level, age, parity, body mass index, country of birth, diabetes mellitus before the pregnancy, certain other pre-pregnancy diseases, previous stillbirth, gestational diabetes mellitus and preeclampsia.

An article describing the study protocol has been published. A pilot study testing complicance of mindfetalness has been published. Data concerning outcome (all recruited women are followed from gestational week 32+0 until delivery) will be exported from the pregnancy register during October 2018.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman with a fetus being at least 25 weeks old (gestational age)
* Having a Swedish personal identity number

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39000 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
An Apgar Score below 7 | Five minutes after birth
  We will use the score assessed in routine care and reported to the Pregnancy Register.
Caesarian section | At delivery
  We will use the information in the Pregnancy Register. The responsible health-care professionals clasify the mode of delivery and report it to the register. The register is population-based and covers by and large every birth in the region at the time.
Induction of Labor | At delivery.
  We will use the information in the Pregnancy Register. The responsible health-care professionals clasify the mode of delivery and report it to the register. The register is population-based and covers by and large every birth in the region at the time.

SECONDARY OUTCOMES:
Visit to health care due to worry about decrease in fetal movements | Pregnancy from week 28
  We will use events registered in the Pregnancy Register.

OTHER OUTCOMES:
An Apgar Score below 4 | Five minutes after birth
  We will use the score assessed in routine care and reported to the Pregnancy Register.
An Apgar Score below 10 | Five minutes after birth
  We will use the score assessed in routine care and reported to the Pregnancy Register.

CONTACTS AND LOCATIONS:
Overall Officials: Ingela Rådestad, PhD, Principal Investigator — Sophiahemmet University
Locations (1):
- Stockholm region, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malm MC, Radestad I, Rubertsson C, Hildingsson I, Lindgren H. Women's experiences of two different self-assessment methods for monitoring fetal movements in full-term pregnancy--a crossover trial. BMC Pregnancy Childbirth. 2014 Oct 7;14:349. doi: 10.1186/1471-2393-14-349. PMID 25288075
- [Background] Radestad I. Strengthening mindfetalness. Sex Reprod Healthc. 2012 Jun;3(2):59-60. doi: 10.1016/j.srhc.2012.01.002. Epub 2012 Jan 27. PMID 22578751
- [Background] Radestad I, Akselsson A, Georgsson S, Lindgren H, Pettersson K, Steineck G. Rationale, study protocol and the cluster randomization process in a controlled trial including 40,000 women investigating the effects of mindfetalness. Sex Reprod Healthc. 2016 Dec;10:56-61. doi: 10.1016/j.srhc.2016.10.004. Epub 2016 Oct 26. PMID 27938874
- [Background] Akselsson A, Georgsson S, Lindgren H, Pettersson K, Radestad I. Women's attitudes, experiences and compliance concerning the use of Mindfetalness- a method for systematic observation of fetal movements in late pregnancy. BMC Pregnancy Childbirth. 2017 Oct 16;17(1):359. doi: 10.1186/s12884-017-1548-5. PMID 29037234
- [Result] Akselsson A, Lindgren H, Georgsson S, Pettersson K, Steineck G, Skokic V, Radestad I. Mindfetalness to increase women's awareness of fetal movements and pregnancy outcomes: a cluster-randomised controlled trial including 39 865 women. BJOG. 2020 Jun;127(7):829-837. doi: 10.1111/1471-0528.16104. Epub 2020 Feb 8. PMID 31971325
- [Derived] Lindgren H, Radestad I, Pettersson K, Skokic V, Akselsson A. Epidural use among women with spontaneous onset of labour - an observational study using data from a cluster-randomised controlled trial. Midwifery. 2021 Dec;103:103156. doi: 10.1016/j.midw.2021.103156. Epub 2021 Sep 30. PMID 34634721
- [Derived] Radestad I, Pettersson K, Lindgren H, Skokic V, Akselsson A. Country of birth, educational level and other predictors of seeking care due to decreased fetal movements: an observational study in Sweden using data from a cluster-randomised controlled trial. BMJ Open. 2021 Jun 25;11(6):e050621. doi: 10.1136/bmjopen-2021-050621. PMID 34172554
- [Derived] Akselsson A, Lindgren H, Skokic V, Radestad I. A decrease in cesarean sections and labor inductions among Swedish women by awareness of fetal movements with the Mindfetalness method. BMC Pregnancy Childbirth. 2020 Oct 1;20(1):577. doi: 10.1186/s12884-020-03268-1. PMID 32998708
- See also: A description of the method in 16 different languages — https://www.mindfetalness.com/

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT02865759/SAP_000.pdf